CLINICAL TRIAL: NCT00205634
Title: Macrolide Antibiotic Therapy for Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BG99-486
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis (CF); Macrolide antiobiotics; airway inflammation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Biaxin ( clarithromycin)

SUMMARY:
The purpose of this study is to evaluate whether Biaxin (clarithromycin) improves sputum abnormalities, lung function, and overall feeling of well-being in people with cystic fibrosis (CF). Biaxin is an antibiotic commonly used for the treatment of respiratory infections in people who do not have CF, and is sometimes used in CF patients as well. Studies done in a disease called diffuse panbronchiolitis (which is similar to CF) and some preliminary studies that have been done in CF patients suggest that Biaxin might have a beneficial effect on CF sputum in ways unrelated to its antibiotic activity.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CF
* ability to reliably perform spirometry
* FEV1 of 30% predicted at the time of screening

Exclusion Criteria:

* Mycobacterium in a sputum culture ever recorded
* a respiratory exacerbation requiring IV antibiotics in the 60 days prior
* used a investigational drug or device in the 60 days prior
* significant (>30ml) of hemoptysis in the past year
* require oxygen or have significant liver or renal disease

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2000-12 (Actual); Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Testing - FEV1
Quality of Life

SECONDARY OUTCOMES:
decrease in neutrophil-dominated airway inflammation
decrease in Pseudomonas alginate production in vitro and in the airway

CONTACTS AND LOCATIONS:
Overall Officials: Bruce K Rubin, MEngr,MD,MBA, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States